CLINICAL TRIAL: NCT04905914
Title: A Phase 1/2a, Open-Label, Safety, Pharmacokinetic, And Preliminary Efficacy Study Of Oral ATRN-119 In Patients With Advanced Solid Tumors
Brief Title: Study Of ATRN-119 In Patients With Advanced Solid Tumors
Acronym: ABOYA-119
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AR-276-01
Record Dates: First submitted 2021-05-17; First posted 2021-05-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: 3+3 Dose escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- 50mg ATRN-119 (Experimental): Once daily oral administration.
  Interventions: Drug: ATRN-119
- 100mg ATRN-119 (Experimental): Once daily oral administration.
  Interventions: Drug: ATRN-119
- 200mg ATRN-119 (Experimental): Once daily oral administration.
  Interventions: Drug: ATRN-119
- 350mg ATRN-119 (Experimental): Once daily oral administration.
  Interventions: Drug: ATRN-119
- 400mg ATRN-119 (Experimental): Twice daily oral administration.
  Interventions: Drug: ATRN-119
- 1100mg ATRN-119 (Experimental): Once daily oral administration
  Interventions: Drug: ATRN-119
- 1300mg ATRN-119 (Experimental): Once daily oral administration
  Interventions: Drug: ATRN-119
- 1500mg ATRN-119 (Experimental): Once daily oral administration
  Interventions: Drug: ATRN-119
- 650mg ATRN-119 (Experimental): Twice daily oral administration.
  Interventions: Drug: ATRN-119
- 750mg ATRN-119 (Experimental): Twice daily oral administration.
  Interventions: Drug: ATRN-119
- 550mg ATRN-119 (Experimental): Once or twice daily oral administration
  Interventions: Drug: ATRN-119
- 800 mg ATRN-119 (Experimental): Once daily oral administration
  Interventions: Drug: ATRN-119

INTERVENTIONS:
Drug: ATRN-119 — ATRN-119 is a capsule formulation that will be supplied as 50 mg and 100 mg capsules packed in sealed plastic bottles (n=30) and dispensed by the site pharmacist in combinations to provide the appropriate dose.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of ATRN-119 through the performance of a Phase 1/2a, open-label, safety, PK, and preliminary efficacy study of oral ATRN-119 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* DNA damage response (DDR) mutations documented in the past medical record or confirmed during the screening period.
* Measurable disease defined by RECIST 1.1.
* Life expectancy ≥ 3 months.
* Subject must be capable of oral administration of study medication.

Exclusion Criteria:

* Patient has had a cytotoxic chemotherapy, immunotherapy, radiotherapy or other targeted therapies within 4 weeks.
* Surgical procedure performed within 7 days prior to first scheduled dose of ATRN-119.
* Concomitant treatment with strong inhibitors or inducers of CYP3A4 and CYP2D6.
* Known human immunodeficiency virus infection (HIV).
* Subjects with active viral or bacterial infections and/or receiving systemic antibiotics or anti-viral medications.
* Current or past diagnosis of leukemia within the past 5 years.
* Prior radiotherapy at the target lesion unless there is evidence of disease progression.
* Known CNS metastases or clinical evidence of CNS involvement that is not stable for previous 1 month by radiology documentation (magnetic resonance imaging [MRI] brain).
* History of non-malignant gastronintestinal (GI) bleeding, gastric stress ulcerations, or peptic ulcer disease within the past 3-months.
* Patient has uncontrolled hypertension at time of enrollment.
* Complete left bundle branch block (LBBB), bifascicular block (right bundle branch block [RBBB] with either left anterior hemiblock or left posterior hemiblock).
* Any clinically significant ST segment and/or T-wave abnormalities.
* Myocardial infarction or unstable angina pectoris within 6 months prior to starting study medication.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) will be collected and evaluated based on summary statistics | Day 1 to Day 28
  Treatment-emergent AEs (TEAEs) will be collected and Clinical Laboratory Evaluations will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Miller, RN BSN, Study Director — Aprea Therapeutics Inc
Locations (7):
- United States (7):
  - Yale Cancer Center, New Haven, Connecticut
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Jordan Center for Gynecologic Oncology at Penn Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - NEXT- Oncology Dallas, Irving, Texas
  - NEXT Oncology- San Antonio, San Antonio, Texas
  - NEXT Oncology- Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No